CLINICAL TRIAL: NCT00333073
Title: Effectiveness and Safety of Bulkamid® as Bulking Agent for the Treatment of Female Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contura (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONSUI-EU02
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2013-07

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; Bulkamid
MeSH Terms: conditions — Urinary Incontinence

ARMS (1):
- Bulkamid (Experimental): Submucosal injection of Bulkamid into urethra
  Interventions: Device: Bulkamid

INTERVENTIONS:
Device: Bulkamid — initial injection with option for second (if required)

SUMMARY:
To assess effectiveness of Bulkamid® injection in females suffering from stress or mixed (stress and urge) urinary incontinence after 12 months follow up period

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Symptomatic stress or mixed urinary incontinence for at least 12 months
* Having at least 1 incontinence episode per day over three days

Exclusion Criteria:

* Regular or intermittent users of an urethral catheter
* Pregnant women
* Suffer from severe allergies or anaphylaxis
* Suffer from autoimmune diseases or any unstable or sever cardio-vascular disease
* History of any cancer within the last 5 years
* Previous surgery for the treatment of urinary incontinence, including bulking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-03; Primary Completion 2008-10 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Subjective responder rate after 12 months follow-up | 12 months

SECONDARY OUTCOMES:
ICIQ | Baseline, treatment, 1-, 6-, 12- and 24-months
24 hour urine leakage | Baseline, treatment, 1-, 6-, 12- and 24-months
daily incidence of incontinence episodes | Baseline, treatment, 1-, 6-, 12- and 24-months
Qol | Baseline, treatment, 1-, 6-, 12- and 24-months

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Lose, Prof., MD, Principal Investigator — KAS Glostrup
Locations (10):
- Denmark (2):
  - Skejby Sygehus, Aarhus
  - KAS Glostrup, Glostrup Municipality
- Helsinki University Central Hospital, Helsinki, Finland
- DRK Gemeinnützige Krankenhaus Gmbh, Chemnitz, Germany
- Sweden (2):
  - Karolinska Institutet, Stockholm
  - Södersjukhuset, Stockholm
- United Kingdom (4):
  - Worthing Hospital, Worthing, West Sussex
  - Birmingham Women´s Hospital, Birmingham
  - University Hospital of Hartlepool, Hartlepool
  - St. George´s Hospital, London

REFERENCES:
- See also: Bulkamid Website — http://www.bulkamid.com/